CLINICAL TRIAL: NCT05456035
Title: Social Cognitive Training to Enhance the Efficacy of CBT forDepression in Youth: A Developmental Approach (R33)
Brief Title: CBT Enhanced With Social Cognitive Training vs. CBT Only With Depressed Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Garber, Professor of Psychology and Human Development, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R33MH115125 (NIH); R33MH115125-03 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Depression
Keywords: Depression; Adolescents; Cognitive behavior therapy
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The study has two intervention arms: (1) CBTSCT is cognitive behavioral therapy enhanced with training in social cognitive abilities (e.g., social perspective taking),and (2) CBT only is cognitive behavioral therapy without the additional SCT training component. Adolescents are randomized to either condition.
Who Masked: Outcomes Assessor
Masking Description: The individuals who conduct the assessments of the outcome measures will be unaware of to which condition the participant was randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy plus social cognitive training (CBTSCT) (Experimental): The cognitive behavioral therapy is based on Beck's cognitive therapy model for the treatment of depression. We will conduct individual therapy with depressed adolescents using modules from the Coping with Stress manual used in other depression treatment studies with adolescents. In addition, therapists will teach teens explicitly about theory of mind and social perspective taking during each session and will use examples from the teen's own life to help them learn the skills.
  Interventions: Behavioral: Cognitive behavioral therapy plus social cognitive training (CBTSCT)
- Cognitive behavioral therapy (CBT) (Active Comparator): The cognitive behavioral therapy is based on Beck's cognitive therapy model for the treatment of depression. Therapists will conduct individual therapy sessions with depressed adolescents using modules from the Coping with Stress manual. Social cognitive training will not be provided to teens in this condition.
  Interventions: Behavioral: Cognitive behavioral therapy plus social cognitive training (CBTSCT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy plus social cognitive training (CBTSCT) — The study has two intervention arms to which depressed adolescents will be randomized: (1) CBTSCT is cognitive behavioral therapy enhanced with training in social cognitive abilities (e.g., social perspective taking), and (2) CBT only is cognitive behavioral therapy without the additional social cognitive training component.
  Other Names: Cognitive behavioral therapy (CBT)

SUMMARY:
Depression in youth is a serious public health concern for which more personalized treatments are needed. This randomized controlled trial will test the effect of an intervention aimed at enhancing social cognitive capacities (e.g., ability to take another's perspective), thereby making treatment of depression in youth more efficient and effective. Participants in the R33 (N=82) will be youth between ages 13- through 17-years-old currently experiencing depression. Youth will be randomized to either an enhanced CBT intervention that teaches social cognitive skills, particularly social perspective taking and theory of mind (CBTSCT) as compared to CBT only. The primary target is improvement in both social cognitive skills and depressive symptoms at post-treatment and at a 6-month follow-up.

DETAILED DESCRIPTION:
Depression in adolescents is a recurrent and impairing disorder. Although some treatments have shown modest effects in children and adolescents (e.g., cognitive behavioral therapy - CBT), there remains a critical need to build upon these therapies to reach even more youths with depression. One variable hypothesized to affect children's interpersonal relationships is their level of social cognitive development on abilities particularly relevant to social functioning and CBT (e.g., social perspective taking; theory of mind). This RCT will test the efficacy of an intervention aimed at increasing children's social cognitive (SC) abilities. Adolescents (ages 13-17; N=82) with depression diagnoses or clinical levels of depressive symptoms (PHQ9 >15) will be randomized to either the social cognitive training enhanced CBT (CBTSCT) or CBT only. In the R33 RCT, investigators will conduct a trial aimed at replicating the results of the R61 with a new sample of 82 youth (ages 13-17) randomized to CBTSCT or CBT only. Youth will be evaluated regarding their social cognitive abilities (i.e., theory of mind), level of depressive symptoms, and social functioning at baseline, post-treatment, and at a 6-month follow-up. Finally, investigators will test if increases in social cognitive abilities partially accounted for the relation between treatment condition and decreases in depression. If the CBTSCT intervention significantly improves participants' social cognitive abilities and decreases depressive symptoms, then this will provide therapists with a more efficient and personalized treatment of depression in youth.

ELIGIBILITY:
Inclusion Criteria:

1. Participants ages 13- through 17-years-old
2. Youth must have a diagnosis of a current depressive disorder (e.g., major depressive episode; persistent depressive disorder) or a score on the Patient Health Questionnaire (PHQ9) > 15

Exclusion Criteria:

* ever met criteria for a diagnosis of bipolar disorder, schizophrenia, autism, or conduct disorder
* current alcohol or substance use disorder with significant impairment
* imminent risk of suicide
* reading level < 4th grade

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Faux Pas Recognition Test | after 12 weeks
  Faux Pas Recognition test (FPRT) measures the ability to identify and explain faux pas situations where a character unintentionally insults another person due to lack of knowledge about some key feature of the other character. FPRT contains 8 Faux Pas and 8 control stories without a faux pas. Stories are followed by 8 questions. Higher scores mean better theory of mind.
Children's Depression Rating Scale-Revised | after 12 weeks
  In the R33 RCT, depression will be another primary outcome measured with the CDRS-R, which is a clinical interview with the parent and teen separately, about the youth's depressive symptoms during the last two weeks. Higher scores mean more depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Judy Garber, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No